CLINICAL TRIAL: NCT01755416
Title: Phase 1 Study of Medtronic Closed Loop Device With ePID Algorithm and Enlite Sensors on Adjuvant Therapy With Insulin and Liraglutide to Minimize Post-prandial Hyperglycemia
Brief Title: Liraglutide Versus Insulin Mono-therapy in the Closed Loop Setting
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Rubina Heptulla, Division Chief of Pediatric Endocrinology, Albert Einstein College of Medicine
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2012-503
Record Dates: First submitted 2012-11-21; First posted 2012-12-24 (Estimated); Results first posted 2018-08-21 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 diabetes; closed loop; artificial pancreas; insulin; victoza; liraglutide
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance | interventions — Insulin; Insulin Aspart; Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- Closed loop with sensor and Insulin (Placebo Comparator): subject will be on the closed loop device with enlite sensors for about 27 hours. They will not be on any study medication and will be on insulin alone.
  Interventions: Drug: Closed loop with sensor and Insulin
- Closed loop with sensor, Insulin and Liraglutide (Active Comparator): Subject will be on the closed loop device with enlite sensors for about 27 hours. In addition to being on insulin, they would take a single injection of 1.2 mg of Liraglutide subcutaneously before dinner, on Day 1.
  Interventions: Drug: Closed loop with sensor, Insulin and Liraglutide

INTERVENTIONS:
Drug: Closed loop with sensor and Insulin — Subject will be on the closed loop device with enlite sensors for about 27 hours. They will not be on any study medication and will be on insulin alone.
  Other Names: Novolog
  Arms: Closed loop with sensor and Insulin
Drug: Closed loop with sensor, Insulin and Liraglutide — In this study visit the subject will be on the closed loop device with enlite sensors for about 27 hours. In addition to being on insulin, they would take a single injection of 1.2 mg of Liraglutide subcutaneously before dinner on Day 1.
  Other Names: Victoza
  Arms: Closed loop with sensor, Insulin and Liraglutide

SUMMARY:
Hypothesis: In type 1 diabetes mellitus, in the setting of a closed loop glucose control system: adjunctive therapy with Liraglutide will afford better post-prandial glycemic excursions than insulin mono-therapy.

Specific Aim: To determine if post-prandial glucose excursions are lowered with the addition of Liraglutide compared to insulin mono-therapy.

Study Design: This is a randomized open labeled crossover design trial comparing adjuvant Liraglutide and insulin Vs. insulin mono-therapy using the ePID closed-loop system for insulin delivery.

DETAILED DESCRIPTION:
After the screening visit, subjects will be randomized to come for two overnight visits. Study A- the subjects will be on the closed loop device with Novolog rapid acting insulin. In Study B- in addition to insulin the subjects will take a one time sub cutaneous injection of 1.2 mg of Victoza before dinner on Day 1. Both visits will last for approximately 30 hours and the subjects will be managed by the closed loop device for approximately 25 hours.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years and less than 40 years
* Have had diabetes for at least 1 year, and in good control (HbA1C < 8.5 %)
* Be on continuous subcutaneous insulin infusion using an insulin pump
* Menstruating women must have negative pregnancy test.
* Hemoglobin (Hb) > 12 g/dL
* Either is not treated with or has been on a stable treatment regimen with any of the following medications for a minimum of 3 months prior to Screening:

  a. Oral contraceptives (female subjects)b. Antihypertensive agents c. Lipid-lowering agents d. Thyroid replacement therapy e. Antidepressant agents
* For female subjects:a. Not breastfeeding b. Negative pregnancy test result (human chorionic gonadotropin, beta subunit [βhCG])at Screening c. If of childbearing potential, must practice and be willing to continue to practice appropriate birth control (defined as at least one method which results in a low failure rate, i.e., less than 1% per year, when used consistently and correctly, such as implants, injectable's, hormonal contraceptives, some intrauterine contraceptive devices, sexual abstinence, tubal ligation or occlusion, or a vasectomized partner)during the entire duration of the study and must not be planning to conceive
* Should not have any alcohol or drug dependency as assessed by CRAFFT questionnaire.

Exclusion Criteria:

* Any chronic disease (leukemia, asthma, inflammatory bowel disease, cystic fibrosis, juvenile rheumatoid arthritis, etc., that directly, or as a result of treatment, directly or indirectly affect glucose homeostasis
* Hemoglobin less than 12 g/dl
* Positive pregnancy test in menstruating young women
* Evidence or history of chemical abuse
* HbA1c > 8.5 %
* Weight less than 50 Kg
* History of gastro paresis and on medications that alter gastric emptying
* History of Pancreatitis and impaired renal function
* Hypoglycemic unawareness
* History of sensitivity to 5-HT3 receptor antagonists
* History of QT prolongation or any known cardio-vascular disease
* Concomitant use of both Acetaminophen and vitamin C
* Patients on glucocorticoid therapy
* Known allergy to Liraglutide
* Personal or family history of elevated calcitonin, calcitonin >100 ng/L, medullary thyroid carcinoma or in patients with Multiple Endocrine Neoplasia (MEN) syndrome type 2.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2013-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rubina A Heptulla, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine West Campus CRC, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 20 participants were screened. However only 18 participants were enrolled into the study. Of these 15 participants completed both study visits. Patients were recruited from diabetes clinics, via fliers, and online postings on clinical trial sites.
Groups:
- Closed Loop/Insulin First,Then Closed Loop/Insulin/Liraglutide: Participants underwent Closed Loop with Insulin first, as a continuous subcutaneous infusion for 2 days. Then they underwent the closed loop with Insulin and Liraglutide; insulin as a continuous subcutaneous infusion and liraglutide as a single daily subcutaneous injection of 1.2 mg for the next 2 days. Each visit is 10 days apart.
- Closed Loop/Insulin/Liraglutide First,Then Closed Loop/Insulin: Participants underwent Closed Loop with Insulin and Liraglutide first, insulin as a continuous subcutaneous infusion and liraglutide as a single daily subcutaneous injection of 1.2 mg for the first 2 days. Then they underwent the closed loop with Insulin alone, as a continuous subcutaneous infusion for the next 2 days. Each visit is 10 days apart.
Period: First Intervention ( Upto 2 Days)
Arm/Group | Closed Loop/Insulin First,Then Closed Loop/Insulin/Liraglutide | Closed Loop/Insulin/Liraglutide First,Then Closed Loop/Insulin
Started | 9 | 9
Completed | 8 | 7
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 2
Period: Second Intervention (Upto 2 Days)
Arm/Group | Closed Loop/Insulin First,Then Closed Loop/Insulin/Liraglutide | Closed Loop/Insulin/Liraglutide First,Then Closed Loop/Insulin
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants who were randomized to receive either Closed Loop/Insulin subcutaneously or Closed Loop /Insulin/Liraglutide; 1.2 mg of Liraglutide subcutaneously as a single daily injection and insulin as a continuous subcutaneous infusion
Arm/Group | All Study Participants
Number analyzed (Participants) | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 26 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 8
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Blood Glucose Measures in Subjects on Closed Loop With Insulin and Liraglutide, Compared to the Closed Loop With Insulin Alone
Description: Measure of targeted blood glucose levels in the Closed Loop setting in the treatment arm, with the addition of Liraglutide compared to insulin monotherapy (continuous subcutaneous insulin infusion)
Time Frame: 0-1500 min
Measure: Mean (Standard Deviation); unit: mg/dl
Groups:
- Closed Loop/Insulin: Participants on Closed Loop with Insulin as a continuous subcutaneous infusion for 2 days
- Closed Loop/Insulin/Liraglutide: Participants on Closed Loop with Insulin and Liraglutide, insulin as a continuous subcutaneous infusion and Liraglutide as a single daily subcutaneous injection of 1.2 mg for 2 days
Arm/Group | Closed Loop/Insulin | Closed Loop/Insulin/Liraglutide
Number analyzed (Participants) | 15 | 15
mg/dl | 159.7 (50.9) | 144.6 (36.3)

ADVERSE EVENTS:
Time Frame: 12 Months
Arm/Group | Closed Loop/Insulin | Closed Loop/Insulin/Liraglutide
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No